CLINICAL TRIAL: NCT06576739
Title: Efficacy and Duration of Chiropractic Spinal Manipulation in Chronic Back Pain With the Inclusion of Vitamins B6, B9, and B12: A Pilot, Placebo-Controlled, Double Blinded Randomized Controlled Trial
Brief Title: B Vitamin Supplementation to Chiropractic Management of Chronic LBP: Pilot Clinical Trial (VCLBP)
Acronym: VCLBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western States (Other)
Responsible Party: Principal Investigator, Anthony Rosner, Research Director, University of Western States
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP Vitamin LBP
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Pilot, Placebo-Controlled, Double Blinded, Randomized Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient, Provider, and Statistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin Administration (Experimental): Vitamins B6, B12, and folic acid will be administered orally between 8:30 am - 10:30 am on day of chiropractic manipulation Chiropractic intervention will be applied Number of patients in arm anticipated: 30
  Interventions: Procedure: Spinal Manipulation
- Placebo Administration (Placebo Comparator): Placebo pills equal in number and appearance to the B vitamins will be administered orally between 8:30 am - 10:30 am on day of chiropractic intervention Chiropractic intervention will be applied Number of patients in arm anticipated: 30
  Interventions: Procedure: Spinal Manipulation

INTERVENTIONS:
Procedure: Spinal Manipulation — Daily administration of combination of vitamin B6,,vitamin B12, and folic acid
  Other Names: B vitamin supplementation

SUMMARY:
The purpose of this investigation is to assess the effects of a combination of B vitamins (B6 [pyridoxine],, B9 [folate], and B12 [cyanocobalamin] upon the efficacy and duration of spinal manipulation in its treatment of chronic low back pain. Outcome measures over a 12-week period include disability (the Oswestry Disability Index), pain (the Quadruple Visual Analog Scale), and quality of life (Short Form 36 Scale). A total of 60 patients are to be recruited by a single practicing chiropractor who will randomize consenting patients into two groups of 30, one of which will take 3 tablets of the Standard Process folic acid B12 and one tablet of Standard Process B6 Niacinamide between 8:30 - 10:30 am each day and the other 4 tablets of placebo fabricated by Standard Process. Both groups will receive treatments from their chiropractor in the manner they would normally experience as patients. Outcomes will be measured 2 weeks prior to commencing the protocol (baseline), at baseline, immediately upon commencing the protocol, and at one, 2, and 3 months following.. Hypotheses are as follows:

HO: Differences in the Oswestry Disability Index (primary outcome) between the experimental and placebo groups will not be clinically and statistically significant at 3 months of treatment.

HA: Differences in the Oswestry Disability Index (primary outcome) between the experimental and placebo groups will be clinically and statistically significant at 3 months of treatment.

Secondary outcomes will be evaluated in the same manner.

DETAILED DESCRIPTION:
As groundwork for a randomized controlled trial, this investigation proposes a pilot study in the management of chronic inflammatory low back pain in patient cohorts under the routine chiropractic care of a given physician, at the same time ingesting daily doses at the same hour each day over a period of 3 months after being randomized to either placebo or a combination of vitamins B6, B9 (folate), and B12 in respective doses of 50 mg, 1.2 mg, and 18 mcg. The targeted number of patients is 48, with 60 recruited to account for dropouts. Inclusion criteria will be (i) ages 18-60, and (ii) chronic inflammatory low back pain experienced constantly or frequently for at least 3 months and screened according to the criteria shown above in TABLE 1, omitting the age criterion. Exclusion criteria will include (i) taking of any antacids, digestive medications, or corticosteroids within the past 30 days, (ii) taking of any of the vitamins B6, B9 (folate), or B12 or a multivitamin capsule containing any of these vitamins within the past 15 days, (iii) not having diagnosed with impaired renal function or chronic kidney disease,1, 2 (iv) currently undergoing therapy for depression or suicidal ideation, (v) the presence of any red flag conditions, such as bowel, bladder, sexual or other dysfunctions; (vi) current involvement with medico-legal proceeding such as workers' compensation claims; or (vii) pregnancy.

Expected outcomes monitored at 2 weeks prior to baseline, at baseline before and after treatment, and at 1, 2, and 3 months after the commencement of treatment will include the Oswestry Disability Index (ODI) as the primary outcome. Secondary outcomes will include (i) the Quadruple Visual Analog Scale (VAS), and (ii) the Short Form Health Survey. Both within-group and between-group comparisons will be made for each chiropractic cohort. A VAS change in the order of 2 units (20 mm) or greater is considered to be of clinical significance in a population low back pain sufferers,3 4 while the minimum clinically important difference for the ODI has been shown to be 6 points, corresponding to 12 percentage points.5, 6

Sample size was previously determined to be 60 participants in treatment and control groups assuming 80% power and α of 0.05 to yield change of ODI of 9 points and SD of 16.29 as previously described.7This is divided among the three participating chiropractors.

For this pilot study, a single chiropractor with a patient cohort of n = 60, randomized into two groups of a minimum 24 each (allowing for dropouts) allocated to placebo or vitamin regimen, will be chosen. We realize that other components in people's diets have ability to produce or suppress inflammation, but our thinking is that (1) the randomization has the capacity to compensate for these effects, and (2) the vitamin supplements have shown a specific ability to significantly suppress homocysteine as a primary inflammatory agent.

After patients agree to participate, they will be further screened with a questionnaire to determine the nature of their back pain, checking off the characteristics that apply to them (Table 1).

TABLE 1: Back pain characteristics

COLUMN A:

* Gradual onset developed over 3+ months
* Pain improves with exercise
* Pain does not improve with rest
* Morning stiffness more than 30 minutes
* Pain at night may wake you up, especially 2nd half of night

COLUMN B: :

* Onset after an event, such as an accident, fall, etc.
* Pain often improves with rest
* Morning stiffness that improves in a few minutes

Patients checking at least 4 of the items in Column A and no more than one in Column B will be further admitted in the effort to obtain as large a sample of inflammatory back pain patients as possible. These participants will be asked to provide written consent to participate in the study after they have read through and understood this document. The participant will be coded (masked) with a 3-digit number that will remain with that individual throughout the duration of the study. The number will be put into a computer to randomize the individual into one of two groups labeled A and B, one of which will be assigned to take the vitamin pills and the other to take an equal number of placebo pills that have identical appearances. Active and placebo preparations will be labeled X and Y upon distribution so as to blind treating doctors as well as patients. The participant will be given questionnaires to assess pain, disability, and quality of life, and then the individual will be asked to return in 2 weeks and complete the questionnaires once again. At this time the participant will receive the chiropractic care that the and his or her doctor find to be best suited to that person's back pain. At the conclusion of the patient's visit, which should last no longer than 20 minutes, the participant will be given 1 pill of Standard Process B6 Niacinamide (#1280) and 3 pills of Standard Process Folic Acid B12 (#4410) or 4 placebo pills (1 matching #1280 lacking the vitamins + 3 matching #4410 lacking the vitamins) depending upon which group the individual have been assigned and told to take the 4 pills once a day between 8:30 am - 10:30 am each day and keep a written diary to that effect, noting any days that were missed and unexpected health events as well . The patient will also complete the same questionnaires a third time at the conclusion of this visit and then continue to visit his or her chiropractor as often as the individual and his or her doctor believe is warranted. Patients will complete the three questionnaires 30, 60, and 90 days after the commencement of treatment, at which time the taking of pills and the study is concluded. At that time, the participant will asked which of the groups A or B the individual believes that he or she was assigned to. When the final data is collated and analyzed, the participant will be informed of the results of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 Chronic inflammatory low back pain experienced constantly or frequently for at least 3 months

Exclusion Criteria:

* Taking any of the vitamins B6, B12, or folic acid or a multivitamin capsule containing any of these vitamins within the past 15 days Not having been diagnosed with impaired renal function or impaired kidney disease Currently undergoing therapy for depression or suicidal ideation Presence of any red flag conditions, such as bowel, bladder, sexual or other dysfunctions Current involvement with medico-legal proceeding such as workers' compensation or claims Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 weeks prior to basel;ne, at baseline; time 0 immediately after first chiropractic treatment; 30 days, 60 days, and 90 days immediately after chiropractic treatment
  Validated paper questionnaire

SECONDARY OUTCOMES:
Quadruple Visual Analog Scale | 2 weeks prior to baseline; at baseline; time 0 immediately after first chiropractic treatment; 30 days, 60 days, amnd 90 days after chiropractic treatment
  Validated paper questionnaire
Short Form (SF-36) Health Survey | 2 weeks prior to baseline; at baseline; time 0 immediately after first chiropractic treatment; 30 days, 60 days, and 90 days after chiropractic treatment
  Validated paper questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Western States, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Collated data statistical analysis, informed consent form will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anticipated June 2025
Access Criteria: Certified professional/individual with institutional affilitation

REFERENCES:
- [Result] Goertz CM, Long CR, Vining RD, Pohlman KA, Walter J, Coulter I. Effect of Usual Medical Care Plus Chiropractic Care vs Usual Medical Care Alone on Pain and Disability Among US Service Members With Low Back Pain: A Comparative Effectiveness Clinical Trial. JAMA Netw Open. 2018 May 18;1(1):e180105. doi: 10.1001/jamanetworkopen.2018.0105. PMID 30646047
- [Result] Rosner AL, Conable KM, Edelmann T. Influence of foot orthotics upon duration of effects of spinal manipulation in chronic back pain patients: a randomized clinical trial. J Manipulative Physiol Ther. 2014 Feb;37(2):124-40. doi: 10.1016/j.jmpt.2013.11.003. Epub 2014 Jan 10. PMID 24412249
- [Result] Pezzini A, Del Zotto E, Archetti S, Negrini R, Bani P, Albertini A, Grassi M, Assanelli D, Gasparotti R, Vignolo LA, Magoni M, Padovani A. Plasma homocysteine concentration, C677T MTHFR genotype, and 844ins68bp CBS genotype in young adults with spontaneous cervical artery dissection and atherothrombotic stroke. Stroke. 2002 Mar;33(3):664-9. doi: 10.1161/hs0302.103625. PMID 11872884
- [Result] Poddar R, Sivasubramanian N, DiBello PM, Robinson K, Jacobsen DW. Homocysteine induces expression and secretion of monocyte chemoattractant protein-1 and interleukin-8 in human aortic endothelial cells: implications for vascular disease. Circulation. 2001 Jun 5;103(22):2717-23. doi: 10.1161/01.cir.103.22.2717. PMID 11390343
- [Result] Dangour AD, Breeze E, Clarke R, Shetty PS, Uauy R, Fletcher AE. Plasma homocysteine, but not folate or vitamin B-12, predicts mortality in older people in the United Kingdom. J Nutr. 2008 Jun;138(6):1121-8. doi: 10.1093/jn/138.6.1121. PMID 18492844
- [Result] Tucker KL, Qiao N, Scott T, Rosenberg I, Spiro A 3rd. High homocysteine and low B vitamins predict cognitive decline in aging men: the Veterans Affairs Normative Aging Study. Am J Clin Nutr. 2005 Sep;82(3):627-35. doi: 10.1093/ajcn.82.3.627. PMID 16155277
- [Result] Smith AD, Smith SM, de Jager CA, Whitbread P, Johnston C, Agacinski G, Oulhaj A, Bradley KM, Jacoby R, Refsum H. Homocysteine-lowering by B vitamins slows the rate of accelerated brain atrophy in mild cognitive impairment: a randomized controlled trial. PLoS One. 2010 Sep 8;5(9):e12244. doi: 10.1371/journal.pone.0012244. PMID 20838622
- [Result] Homocysteine Lowering Trialists' Collaboration. Dose-dependent effects of folic acid on blood concentrations of homocysteine: a meta-analysis of the randomized trials. Am J Clin Nutr. 2005 Oct;82(4):806-12. doi: 10.1093/ajcn/82.4.806. PMID 16210710
- [Result] Clarke R, Halsey J, Lewington S, Lonn E, Armitage J, Manson JE, Bonaa KH, Spence JD, Nygard O, Jamison R, Gaziano JM, Guarino P, Bennett D, Mir F, Peto R, Collins R; B-Vitamin Treatment Trialists' Collaboration. Effects of lowering homocysteine levels with B vitamins on cardiovascular disease, cancer, and cause-specific mortality: Meta-analysis of 8 randomized trials involving 37 485 individuals. Arch Intern Med. 2010 Oct 11;170(18):1622-31. doi: 10.1001/archinternmed.2010.348. PMID 20937919
- [Result] Mauro GL, Martorana U, Cataldo P, Brancato G, Letizia G. Vitamin B12 in low back pain: a randomised, double-blind, placebo-controlled study. Eur Rev Med Pharmacol Sci. 2000 May-Jun;4(3):53-8. PMID 11558625